CLINICAL TRIAL: NCT04211753
Title: Effectiveness and Security Testing of a Mobile App (B·RIGHT) for Self-managing Emotional Crises in People With Borderline Personality Disorder: A Pragmatic Randomized Controlled Trial
Brief Title: Effectiveness and Security Testing of a Mobile App (B·RIGHT) for Emotional Crisis in Borderline Personality Disorder
Acronym: B·RIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIC 32/16
Record Dates: First submitted 2019-12-19; First posted 2019-12-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline personality disorder; Mobile app; Crisis intervention; Effectiveness; Security
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Therapeutics; Schema Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual plus mobile app (Experimental): Those who will receive naturalistic treatment in outpatient setting and also the mobile app
  Interventions: Behavioral: Treatment as usual (schema therapy); Device: Mobile app
- Treatment as usual (Active Comparator): Those who will receive naturalistic treatment in outpatient setting but not the mobile app
  Interventions: Behavioral: Treatment as usual (schema therapy)

INTERVENTIONS:
Behavioral: Treatment as usual (schema therapy) — weekly group psychotherapy and bimonthly individual psychotherapy
Device: Mobile app — Medical device for crisis intervention
  Arms: Treatment as usual plus mobile app

SUMMARY:
To assess the effectiveness and security of a mobile App (beta version) for self-managing emotional crisis in a pragmatic randomized controlled trial with 80 patients with borderline personality disorder (40 patients with treatment as usual, TAU) versus 40 patients with TAU plus the mobile App)

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) of borderline personalidad disorder (BPD)
* Aged 18-60 yeats old

Exclusion Criteria:

* Comorbidity with mental retardation
* Comorbidity with psychotic disorder
* Comorbidity with antisocial personality
* Comorbidity with autism spectrum disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Number of psychiatric.emergencies and hospitalizations | 9-month
  As reported by computerized clinical charts
smartphone addiction | 9-month
  Severity of smartphone addiction as measured by the Spanish version of the Smartphone Addiction Scale (SAS) (range: 10-60; the higher the score, the more severe the smartphone addiction severity).

CONTACTS AND LOCATIONS:
Overall Officials: Pere Clave, Study Director — Consorci Sanitari del Maresme
Locations (1):
- Consorci Sanitari del Maresme, Mataró, Barcelona, Spain